CLINICAL TRIAL: NCT06316687
Title: Prevalence of Dental Caries in a Group of Egyptian Children and Its Relation to TV and Other Screens Time and Sugar Consumption
Brief Title: Prevalence of Dental Caries in a Group of Egyptian Children
Status: Not yet recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mona Elhadi Elamin, Dr Mona Elhadi Elamin, Cairo University
Other Study IDs: prevalence of dental caries
Record Dates: First submitted 2024-03-12; First posted 2024-03-18 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Prevalence of Dental Caries and Its Relation to Screen Time and Sugar Consumption; Prevalence,Patient
Keywords: prevalence; dental caries; screen time; sugar consumption
MeSH Terms: conditions — Dental Caries | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: questionnaire for food consumption frequency — questionnaire about Food consumption frequency, Screen time , Dental neglect scale
  Other Names: screen time; Dental neglect scale

SUMMARY:
Prevalence of Dental Caries in a group of Egyptian children and its relation to TV and other screens time and sugar consumption (Observational cross-sectional study)

DETAILED DESCRIPTION:
Dental caries, are considered by the World Health Organization as a major public health problem globally, and the most widespread non-communicable disease.

Similar with other conditions that are described as non-communicable diseases (NCDs), dental caries develops as the result of a combination of genetic, physiological, environmental and behavioral factors.

The commonly accepted risk factors for dental caries include dietary habits (e.g., sugary snacks), poor oral hygiene, microbiological factors, and low socioeconomic status.

Watching TV during mealtime has a negative impact on children's dietary quality as it is associated with higher consumption of ultraprocessed foods .

It was found that having the TV on at mealtimes reduces diet quality with more high-fat, high-sugar foods and fewer fruits and vegetables and increased consumption of sugar sweetened beverages.

Overconsumption of sugar has been associated with increased risk of excessive weight gain, dental decay, poor diet quality and nutritional inadequacy in children and adolescents younger than 19 years .

ELIGIBILITY:
Inclusion Criteria:

* 1. A child with mixed dentition aged from 6-8 years old 2. Positive subject acceptance for participation in the study 3. Access to all types of screens 4. Both gender

Exclusion Criteria:

* 1. A child with a dental emergency 2. Child with a psychological problem 3. Child with chronic illness

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: male and female healthy children aged from 6 - 8 years who have access to different types of screens and willing to participate
Sampling Method: Probability Sample
Enrollment: 296 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of dental caries | 1 month
  Visual Inspection and intraoral examination using DMF, def

SECONDARY OUTCOMES:
Dental neglect Dental neglect Dental neglect | 1 month
  Questionnaire, Dental neglect scale (DNS)
Screen time evaluation | 1 month
  The range of time spent by children using screens will be reported daily by parents on weekdays and weekend days for a week
A sugar consumption evaluation | 1 month
  Health Behavior in School-Aged Children Food-Frequency Questionnaire (HBSC-FFQ).

CONTACTS AND LOCATIONS:
Overall Officials: mona El tayeb, master, Principal Investigator — Cairo University
Locations (1):
- Cairo University, Cairo, Al Manial, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
calculating the prevalence of dental caries among Egyptian children using DMF and def, and if there is a relation to screen time and sugar consumption using questionnaires

REFERENCES:
- [Background] Abbass MMS, Mahmoud SA, El Moshy S, Rady D, AbuBakr N, Radwan IA, Ahmed A, Abdou A, Al Jawaldeh A. The prevalence of dental caries among Egyptian children and adolescences and its association with age, socioeconomic status, dietary habits and other risk factors. A cross-sectional study. F1000Res. 2019 Jan 3;8:8. doi: 10.12688/f1000research.17047.1. eCollection 2019. PMID 30854195
- [Background] Yilmaz N, Avci G. Exposure to screen time and dental neglect. J Paediatr Child Health. 2022 Oct;58(10):1855-1861. doi: 10.1111/jpc.16177. Epub 2022 Aug 18. PMID 36181437
- [Background] Madigan S, Browne D, Racine N, Mori C, Tough S. Association Between Screen Time and Children's Performance on a Developmental Screening Test. JAMA Pediatr. 2019 Mar 1;173(3):244-250. doi: 10.1001/jamapediatrics.2018.5056. PMID 30688984
- [Background] Martines RM, Machado PP, Neri DA, Levy RB, Rauber F. Association between watching TV whilst eating and children's consumption of ultraprocessed foods in United Kingdom. Matern Child Nutr. 2019 Oct;15(4):e12819. doi: 10.1111/mcn.12819. Epub 2019 May 23. PMID 30941879
- [Background] Shqair AQ, Pauli LA, Costa VPP, Cenci M, Goettems ML. Screen time, dietary patterns and intake of potentially cariogenic food in children: A systematic review. J Dent. 2019 Jul;86:17-26. doi: 10.1016/j.jdent.2019.06.004. Epub 2019 Jun 19. PMID 31228564